CLINICAL TRIAL: NCT03859713
Title: Optimized Multidisciplinary Treatment Programs for Nonspecific Chronic Low Back Pain
Brief Title: Optimize Low Back Pain
Acronym: OPTIMIZE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Utah (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Julie Fritz, Distinguished Professor, University of Utah
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 00116150
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Low Back Pain; Chronic Pain
Keywords: Physical Therapy; Cognitive Behavioral Therapy; Mindfulness; Adaptive Treatment Regimens
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Physical Therapy Modalities; Cognitive Behavioral Therapy; Mindfulness

STUDY DESIGN:
Intervention Model Description: Our design is a sequential multiple randomization (SMART) study design with 2 treatment phases with a possibility of 2 randomizations per participant.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and clinicians cannot be blind to treatment received. The investigators will remain blind to group assignment and follow-up assessments will be conducted by assessors who are blind to treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PT followed by Switching to CBT in Phase II for nonresponders (Experimental): Phase I treatment is 8 weekly sessions of evidence-based physical therapy (PT). At the 10-week follow-up participants who are non-responders to Phase I PT will switch to 8 weekly sessions of cognitive behavioral therapy (CBT) as Phase II treatment. If participant is a responder to Phase I PT, he or she will receive up to 2 more PT sessions in Phase II of treatment.
  Interventions: Behavioral: Physical Therapy; Behavioral: Cognitive Behavioral Therapy
- PT followed by Mindfulness in Phase II for nonresponders (Experimental): Phase I treatment is 8 weekly sessions of evidence-based physical therapy (PT). At the 10-week follow-up participants who are non-responders to Phase I PT will receive 8 weekly sessions of mindfulness using a mindfulness-oriented recovery enhancement protocol as Phase II treatment. If participant is a responder to Phase I PT, he or she will receive up to 2 more PT sessions in Phase II of treatment.
  Interventions: Behavioral: Physical Therapy; Behavioral: Mindfulness
- CBT followed by Switching to PT in Phase II for nonresponders (Experimental): Phase I treatment is 8 weekly sessions of cognitive behavioral therapy (CBT). At the 10-week follow-up participants who are non-responders to Phase I CBT will switch to 8 weekly sessions of evidence-based physical therapy (PT) as Phase II treatment. If participant is a responder to Phase I CBT, he or she will receive up to 2 more CBT sessions in Phase II of treatment.
  Interventions: Behavioral: Physical Therapy; Behavioral: Cognitive Behavioral Therapy
- CBT followed by Mindfulness in Phase II for nonresponders (Experimental): Phase I treatment is 8 weekly sessions of cognitive behavioral therapy (CBT). At the 10-week follow-up participants who are non-responders to Phase I CBT will switch to 8 weekly sessions of mindfulness using a mindfulness-oriented recovery enhancement protocol as Phase II treatment. If participant is a responder to Phase I CBT, he or she will receive up to 2 more CBT sessions in Phase II of treatment.
  Interventions: Behavioral: Cognitive Behavioral Therapy; Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Physical Therapy — Evidence-based physical therapy provided in 8 individual sessions including patient education, exercise instruction and manual therapy.
  Arms: CBT followed by Switching to PT in Phase II for nonresponders; PT followed by Mindfulness in Phase II for nonresponders; PT followed by Switching to CBT in Phase II for nonresponders
Behavioral: Cognitive Behavioral Therapy — Evidence-based cognitive behavioral therapy provided in 8 individual sessions focused on key components of CBT; 1) identifying and monitoring maladaptive cognitions, 2) developing coping strategies (e.g., distraction, relaxation, etc.), 3) setting and working towards behavioral goals, especially focused on physical activity, and 4) focusing on self-management skills and home instruction
  Arms: CBT followed by Mindfulness in Phase II for nonresponders; CBT followed by Switching to PT in Phase II for nonresponders; PT followed by Switching to CBT in Phase II for nonresponders
Behavioral: Mindfulness — Mindfulness is provided in 8 individual sessions. Focus of sessions is cognitive reappraisal, positive savoring and mindfulness practices.
  Other Names: Mindfulness-Oriented Recovery Enhancement
  Arms: CBT followed by Mindfulness in Phase II for nonresponders; PT followed by Mindfulness in Phase II for nonresponders

SUMMARY:
The objective of this study is to improve health care for patients with chronic LBP and increase the likelihood that patients obtain outcomes that matter most to them. The investigators will accomplish our goal using a sequential multiple randomization (SMART) design comparing the effectiveness of Phase 1 (PT v. CBT) treatments for patients with chronic LBP; and among patient non-responsive to Phase I treatment, compare the effectiveness of Phase II treatments (switching to PT or CBT v. mindfulness). Effectiveness will be based on patient-centered outcomes. Sub-aims will compare main effects of Phase 1 and 2 treatment options and the sequencing effects of different treatment combinations.

DETAILED DESCRIPTION:
The study uses a sequential multiple randomization (SMART) design. The study will compare the effectiveness of common first-line treatments for chronic LBP: PT or CBT. Initial treatment will be 8 weeks duration with re-evaluation at 10-weeks after enrollment to allow time to complete treatment. At the 10-week assessment researchers will examine if the patient has responded to initial treatment using a patient-centered, validated definition of successful response based on 50% improvement in the Oswestry Disability Index (ODI). Patients who are responders to initial treatment will receive up to 2 additional sessions of the same treatment to assist transition to self-management. Non-responders will be re-randomized to a second treatment strategy of either switching to the other initial treatment (i.e., patients receiving PT switch to CBT or vice versa), or mindfulness. The second treatment phase is also 8 weeks in duration. Additional follow-ups occur 26- and 52 weeks after enrollment.

The study has two co-primary outcomes; function and pain. The investigators will use the ODI, a well-validated, reliable and responsive patient-reported measure of LBP-related function recommended by the NIH Back Pain Task Force. The investigators will assess pain intensity with 0-10 ratings ('0' indicating no pain and '10' worst imaginable pain). Separate ratings are made for current, worst and best pain over the past 24 hours with an average computed to represent pain intensity. Secondary outcomes will assess dimensions of quality of life, work and healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 64 years at the time of enrollment.
* Meets NIH Task Force definition of chronic LBP based on two questions: 1) How long has LBP has been an ongoing problem for you? and 2) How often has LBP been an ongoing problem for you over the past 6 months? A response of greater than 3 months to question 1, and "at least half the days in the past 6 months" to question 2 is required to satisfy the NIH definition of chronic LBP.
* Healthcare visit for LBP in the past 90 days.
* At least moderate levels of pain and disability requiring ODI score >24 and pain intensity rating > 4.
* Has access to two-way video technology, such as smartphone, iPad/tablet, or laptop with webcam for telehealth visits.

Exclusion Criteria:

* Evidence of serious pathology as a cause of LBP including neoplasm, inflammatory disease (e.g., ankylosing spondylitis), vertebral osteomyelitis, etc.
* Evidence of a specific spinal pathology as the cause of LBP including spine fracture, spinal stenosis, radiculopathy, etc.
* Knowingly pregnant
* Has received physical therapy for LBP; or CBT or mindfulness for any reason with a provider in prior 90 days
* Currently receiving substance use disorder treatment
* Any lumbar spine surgery in the past year.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 748 (Estimated)
Dates: Start 2019-03-22 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index from baseline to 10 weeks | baseline, 10 weeks
  Back pain specific measure of functional disability to address Aim 1
Change in Oswestry Disability Index from baseline to 52 weeks | baseline, 52 weeks
  Back pain specific measure of functional disability to address Aim 2
Change in Numeric Pain Intensity Rating from baseline to 10 weeks | baseline, 10 weeks
  0-10 numeric rating of pain intensity measured as average of current, best and worst pain ratings in past 24 hours to address Aim 1.
Change in Numeric Pain Intensity Rating from baseline to 52 weeks | baseline, 52 weeks
  0-10 numeric rating of pain intensity measured as average of current, best and worst pain ratings in past 24 hours to address Aim 2.

SECONDARY OUTCOMES:
Health-related Quality of Life | baseline, 10 weeks, 26 weeks, 52 weeks
  PROMIS-29 score assessed as a T-score with mean = 50 and SD = 10
Pain Interference | baseline, 10 weeks, 26 weeks, 52 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Fatigue | baseline, 10 weeks, 26 weeks, 52 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Sleep Disturbance | baseline, 10 weeks, 26 weeks, 52 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Anxiety | baseline, 10 weeks, 26 weeks, 52 weeks
  PROMIS 4-item short form (part of PROMIS-29)assessed as a T-score with mean = 50 and SD = 10
Depression | baseline, 10 weeks, 26 weeks, 52 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Social Role Participation | baseline, 10 weeks, 26 weeks, 52 weeks
  PROMIS 4-item short form (part of PROMIS-29) assessed as a T-score with mean = 50 and SD = 10
Health Care Utilization | baseline, 10 weeks, 26 weeks, 52 weeks
  Utilization of surgery, injections, imaging or other discrete interventions for low back pain
Opioid Utilization | baseline, 10 weeks, 26 weeks, 52 weeks
  Use of opioids for pain management
Treatment Side Effects | 10 weeks, 26 weeks
  Self-reported physical or psychological side effects of study treatments
Treatment Responder | baseline, 10 weeks, 26 weeks, 52 weeks
  Dichotomous outcome based on achieving at least 50% improvement on ODI from baselin score

CONTACTS AND LOCATIONS:
Overall Officials: Julie Fritz, PT, PhD, Principal Investigator — University of Utah
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - Intermountain Health Care, Salt Lake City, Utah
  - The University of Utah Healthcare System, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skolasky RL, Wegener ST, Aaron RV, Ephraim P, Brennan G, Greene T, Lane E, Minick K, Hanley AW, Garland EL, Fritz JM. The OPTIMIZE study: protocol of a pragmatic sequential multiple assessment randomized trial of nonpharmacologic treatment for chronic, nonspecific low back pain. BMC Musculoskelet Disord. 2020 May 11;21(1):293. doi: 10.1186/s12891-020-03324-z. PMID 32393216
- [Derived] Fritz JM, Greene T, Brennan GP, Minick K, Lane E, Wegener ST, Skolasky RL. Characterizing modifications to a comparative effectiveness research study: the OPTIMIZE trial-using the Framework for Reporting Adaptations and Modifications to Evidence-based Interventions (FRAME). Trials. 2023 Feb 23;24(1):137. doi: 10.1186/s13063-023-07150-1. PMID 36823645
- [Derived] Fritz JM, Lane E, Minick KI, Bardsley T, Brennan G, Hunter SJ, McGee T, Rassu FS, Wegener ST, Skolasky RL. Perceptions of Telehealth Physical Therapy Among Patients with Chronic Low Back Pain. Telemed Rep. 2021 Nov 3;2(1):258-263. doi: 10.1089/tmr.2021.0028. eCollection 2021. PMID 34927165